CLINICAL TRIAL: NCT03477292
Title: A Study to Compare 7-days Versus 14 Days of Antibiotics Therapy for Ventilator Associated Pneumonia Due to Drug Resistant Acinetobacter Baumanii
Brief Title: 7-days Versus 14 Days of Antibiotics Therapy for Ventilator Associated Pneumonia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Inderpaul singh, Assistant Professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IEC/82
Record Dates: First submitted 2018-03-20; First posted 2018-03-26 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Ventilator Associated Pneumonia
MeSH Terms: conditions — Pneumonia, Ventilator-Associated

STUDY DESIGN:
Intervention Model Description: Randomized trial
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Long duration of antibiotics (Experimental): 14 days of Colistin
  Interventions: Drug: Duration of antibiotic
- Short duration of antibiotics (Active Comparator): 7 days of Colistin
  Interventions: Drug: Duration of antibiotic

INTERVENTIONS:
Drug: Duration of antibiotic — Duration of antibiotic for treatment of VAP
  Other Names: Colisitin

SUMMARY:
There is evidence that using shorter antibiotic regimens may help in decreasing antimicrobial resistance and reducing drug-related adverse events.6 Moreover, short-course treatments were found to be as effective as longer-course antibiotic treatment.7,8 In a pooled analysis of four randomized trials in VAP comparing shorter versus long duration of antibiotics in the management of VAP, no difference in the mortality was found. We hypothesize that the use of short course of antibiotics in the treatment of VAP due to drug resistant Acinetobacter baumanii (sensitive to carbapenems and/or colistin only) may result in a higher antibiotic-free days and drug related adverse events, in comparison to a longer duration of antibiotics. In this study, we propose to study a 7-day versus 14-day course of antibiotics in patients with drug-resistant Acinetobacter baumanii.

DETAILED DESCRIPTION:
Ventilator-associated pneumonia (VAP) is one of the major causes of morbidity and mortality in the ICU, accounting for 25% of the total infections occurring in this setting and 50% of all antibiotic prescriptions in patients who are mechanically ventilated.1,2 The incidence of VAP depends not only on the type of the institution, the preventive measures and therapeutic approaches that are used, but also on the type of surveillance systems by which incidence is estimated. There are reports of incidence across different settings varying from 1.4 up to 42.8 episodes of VAP/1,000 ventilation-days.2 Patients with VAP have significantly longer ICU and hospital lengths of stay compared with similar patients without VAP.3,4 Consequently, the economic burden of VAP is considerable, leading to significant draining of resources. Even after adjusting for underlying severity of illness, the attributable cost of VAP amounts to several thousands of US dollars per patient.5 There is evidence that using shorter antibiotic regimens may help in decreasing antimicrobial resistance and reducing drug-related adverse events.6 Moreover, short-course treatments were found to be as effective as longer-course antibiotic treatment.7,8 In a pooled analysis of four randomized trials in VAP comparing shorter versus long duration of antibiotics in the management of VAP, no difference in the mortality was found.9 There was an increase in the antibiotic free days in the short course antibiotic arm. There was no difference in the number of relapses of VAP with either modality of treatment.9 In another analysis of six studies with 1088 subjects, there was a higher occurrence of relapses of VAP due to non-lactose fermenting gram negative organism.10 However, there was no difference in the mortality rates.10 The problem with both these meta-analyses was that they did not provide information regarding the outcomes of VAP due to Acinetobacter baumanii.9,10 Also, the short duration strategy included studies that randomized patients to seven to eight days and ten-to fifteen days in the long duration strategy. None of the previous studies has provided information about outcomes of VAP due to Acinetobacter baumanii. In our observation, most of the episodes of VAP in our ICU are due to drug resistant Acinetobacter baumanii. We hypothesize that the use of short course of antibiotics in the treatment of VAP due to drug resistant Acinetobacter baumanii (sensitive to carbapenems and/or colistin only) may result in a higher antibiotic-free days and drug related adverse events, in comparison to a longer duration of antibiotics. In this study, we propose to study a 7-day versus 14-day course of antibiotics in patients with drug-resistant Acinetobacter baumanii.

ELIGIBILITY:
Inclusion Criteria:

(a) Patients who develop ventilator associated pneumonia due to drug-resistant Acinetobacter baumanii; (b) age group of 18 to 75 years

Exclusion Criteria:

(a) VAP due to other organisms; (b) pregnancy; (c) endotracheal or tracheostomy tube aspirate demonstrating growth of drug sensitive Acinetobacter baumanii or an organism other than Acinetobacter baumanii; and, (c) failure to provide informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Relapses of VAP | 28 days
  defined as repetitive clinically and microbiologically documented VAP due to the same pathogen

SECONDARY OUTCOMES:
Duration of mechanical ventilation | 28 days
  (non-invasive and invasive)
ICU and hospital length of stay | 90 days
  Days spent in ICU and hospital
28-day mortality | 28 days
  ICU or hospital mortality
Antibiotic free days | 28 days
  Number of days spent without antibiotics

CONTACTS AND LOCATIONS:
Locations (2):
- India (2):
  - Respiratory ICU, Department of Pulmonary Medicine, PGIMER, Chandigarh, Chandigarh
  - Respiratory ICU, Post Graduate Institue of Medical Education and Research, Chandigarh, Chandigarh

IPD SHARING:
Plan to Share IPD: Undecided
anonymized individual patient information and clinical details will be shared